CLINICAL TRIAL: NCT05958095
Title: Supporting Maternal Mental Health and Emotional Regulation (SuMMER): Assessment of the Clinical Effectiveness of a Mobile Application for Patients With Postpartum Depression
Brief Title: Curio Digital Therapy for the Treatment of Post-partum Depression
Acronym: SuMMER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Healthcare Innovation Technology Lab (Industry)
Collaborators: Curio Digital Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Stan Kachnowski, Chair, Healthcare Innovation Technology Lab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-T-003
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: PostPartum Depression
Keywords: PostPartum depression (PPD), symptoms of PPD, Anxiety, Peri-natal depression, mild-to-moderate depression
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The data of 200 participants will be collected and analyzed for this study. Participants will be selected from a pool of patients who have given birth in the last three months prior to the study start date and been diagnosed with postpartum depression or have experienced depressive symptoms. The study aims to recruit a diverse study cohort across age, race, and SES to reflect the intended user population in the United States.
Who Masked: Participant
Masking Description: Participants are not aware of whether they are receiving the MamaLift Plus interventional device or the digital placebo device. The applications have the same user interface and require a similar amount of time to complete activities. Participants in both arms will receive treatment as usual in addition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MamaLift Plus (Experimental): Principles of Cognitive Behavioral Therapy used to treat PPD with App
  Interventions: Device: MamaLift Plus
- Digital Sham App (Sham Comparator): Content on general mental health and wellbeing topics delivered with sham App
  Interventions: Device: Digital Sham App

INTERVENTIONS:
Device: MamaLift Plus — MamaLift Plus is a digital therapeutic designed to augment usual care and support the treatment of mild-to-moderate postpartum depression (PPD). This mobile-based intervention is grounded on principles of Cognitive Behavioral Therapy (CBT) and Interpersonal Therapy (IPT) and includes key content areas for the treatment management of PPD. It also includes recent developments in acceptance and commitment-based therapies, specifically for the perinatal context.
  Arms: MamaLift Plus
Device: Digital Sham App — The digital sham app delivers content, tips, and suggestion for general wellbeing support.
  Arms: Digital Sham App

SUMMARY:
Primary Objective: Evaluate the clinical effectiveness of the MamaLift Plus app compared to control (digital sham plus treatment as usual) for the management of PPD in the observed population for a period of 9 calendar weeks. It is hypothesized that women who use the MamaLift Plus APP will experience less severe symptoms of depression in post-partum period than comparable women who do not and receive their usual care from health providers.

DETAILED DESCRIPTION:
Women between 18 and 50 years of age who have had a live birth within 3 months prior to study start date and have a diagnosis of mild to moderate PPD. A total of 200 women will be recruited to volunteer in the study with 166 assigned to the intervention arm and 37 assigned to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to read, write and speak English; 3. Participants must provide written informed consent prior to enrollment; 4. Participants must be 18 to 50 years of age at the time of enrollment; 5. Participants must have had a live childbirth <=3 months prior to their enrollment into the study; 6. Participants who have a score of greater than or equal to 13 but not exceeding 19 on the Edinburgh Postnatal Depression Scale (EPDS) during initial screening visit/call; 7. Depression diagnosis needs to be confirmed by licensed behavioral health therapist or medical professional; 8. Participants must answer "0/Never" or "1/Hardly Ever" to the self-harm question on EPDS (Question #10); 9. Participants must be willing to use a mobile app and own an iOS or android enabled mobile phone or device; 10. Participants must have wireless internet connectivity in their home (or have access to internet connectivity) and be willing to connect devices via a Wi-Fi network

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult females who delivered live births in the 3 months prior to study start
Enrollment: 142 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
EPDS Score | 9 week period
  Proportion of women that improve EPDS by >= 4 points at their end of study assessment.
EPDS Score improvement | 9 week period
  Proportion of women that improve EPDS to < 13 points at their end of study assessment

CONTACTS AND LOCATIONS:
Overall Officials: Stan Kachnowski, PhD, Principal Investigator — Healthcare Innovation Technology Lab
Locations (1):
- Healthcare Innovation and Technology Lab, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dixit S, Malladi I, Shankar S, Shah A. Evaluating the Efficacy of MamaLift Plus Digital Therapeutic Mobile App for Postpartum Depression (SuMMER): Randomized, Placebo-Controlled Pivotal Trial. J Med Internet Res. 2025 Jul 1;27:e69050. doi: 10.2196/69050. PMID 40549508